CLINICAL TRIAL: NCT04655313
Title: An Open Label, 4-Week, Phase 2, Maximal Usage Pharmacokinetics and Safety Study of ARQ-151 Cream 0.3% Administered QD in Pediatric Subjects (Ages 6 to 11 Years Old) With Plaque Psoriasis
Brief Title: Maximal Usage Pharmacokinetics and Safety of ARQ-151 in Children With Plaque Psoriasis (ARQ-151-215)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ-151-215
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Psoriasis; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARQ-151 cream 0.3% (Experimental): Open label study of ARQ-151 cream 0.3% applied once daily for 4 weeks
  Interventions: Drug: ARQ-151 cream 0.3%

INTERVENTIONS:
Drug: ARQ-151 cream 0.3% — ARQ-151 cream 0.3% applied to chronic plaque psoriasis lesions once a day for 4 weeks
  Other Names: Topical roflumilast

SUMMARY:
This is a Phase 2, open label, maximal usage PK and safety study of ARQ-151 cream 0.3% in pediatric subjects (ages 6 to 11 years old) with plaque psoriasis:

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of parent(s) or legal guardian, and, if age appropriate, assent by the subject, as required by local laws.
* Males or females, 6 to 11 years old (inclusive).
* Clinical diagnosis of psoriasis vulgaris of at least 2 months duration as determined by the Investigator or through subject interview. Stable disease for the past 3 weeks.
* Psoriasis vulgaris on the face, extremities, trunk, and/or intertriginous areas involving at least 2% of BSA (excluding the scalp, palms, and soles).
* An Investigator Global Assessment of disease severity (IGA) of at least Mild ('2') at Baseline.
* Subject has adequate venous access for PK sampling in areas not involved by plaque psoriasis and not being treated with ARQ-151 (e.g., back of the hands).
* Females of childbearing potential (FOCBP) must have a negative serum pregnancy test at Screening (Visit 1) and a negative urine pregnancy test at Baseline (Visit 2). In addition, sexually active FOCBP must agree to use at least one form of highly effective contraception throughout the duration of the trial and for one week after application of the last dose.
* Females of non-childbearing potential must be pre-menarchal.
* In good health as judged by the Investigator, based on medical history, physical examination, 12-lead electrocardiogram (ECG), serum chemistry labs, hematology values, and urinalysis.
* Subjects and parent(s)/legal guardian(s) are considered reliable and capable of adhering to the Protocol and Visit Schedule, according to the judgment of the Investigator.

Exclusion Criteria:

* Subjects with any serious medical or psychiatric condition or clinically significant laboratory, ECG, vital signs, or physical examination abnormality that would prevent study participation or place the subject at significant risk, as judged by the Investigator.
* Planned initiation or changes to concomitant medication that could, in the opinion of the Investigator, affect psoriasis vulgaris
* Current diagnosis of non-plaque form of psoriasis (e.g., guttate, erythrodermic/exfoliative, palmoplantar only involvement, or pustular psoriasis). Current diagnosis of drug-induced psoriasis.
* Subjects with any condition on the treatment area which, in the opinion of the Investigator, could confound efficacy measurements.
* Subjects who cannot discontinue the use of strong cytochrome P-450 CYP3A4 inducers for 2 weeks prior to Baseline/Day 1and during the study period.
* Subjects who cannot discontinue the use of strong cytochrome P-450 CYP3A4 inhibitors for 2 weeks prior to Baseline/Day 1 and during the study period.
* Subjects who are unwilling to refrain from prolonged sun exposure and from using a tanning bed or other artificial light emitting devices (LEDs) for 4 weeks prior to Baseline/Day 1 and during the study.
* Subjects who cannot discontinue specific systemic therapies and/or topical therapies prior to the Baseline/Day 1 and during the study period according to the protocol.
* Subjects with any infection requiring oral or intravenous administration of antibiotics, antifungal or antiviral agents within 2 weeks prior to Baseline/Day 1.
* Subjects with a CDI-2 (parent report) raw score >20 at Screening/Baseline

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (17):
- United States (15):
  - Arcutis Clinical Site 503, Mountain Brook, Alabama
  - Arcutis Clinical Site 504, Scottsdale, Arizona
  - Arcutis Clinical Site 509, Fountain Valley, California
  - Arcutis Site 518, Los Angeles, California
  - Arcutis Clinical Site 508, Los Angeles, California
  - Arcutis Clinical Site 511, Rancho Santa Margarita, California
  - Arcutis Clinical Site 510, Boca Raton, Florida
  - Arcutis Clinical Site 502, Coral Gables, Florida
  - Arcutis Clinical Site 513, Delray Beach, Florida
  - Arcutis Clinical Site 501, Hialeah, Florida
  - Arcutis Clinical Site 507, Miami, Florida
  - Arcutis Clinical Site 527, West Lafayette, Indiana
  - Arcutis Clinical Site 506, Arlington, Texas
  - Arcutis Clinical Site 519, Frisco, Texas
  - Arcutis Clinical Site 505, Houston, Texas
- Arcutis Clinical Site 521, Toronto, Ontario, Canada
- Arcutis Clinical Site 530, Santo Domingo, Dominican Republic

REFERENCES:
- [Derived] Hebert AA, Guide SV, Groysman V, Gonzalez ME, Blanco D, Laquer V, Seal MS, Thurston A, Krupa D, Snyder S, Burnett P, Chu DH, Berk DR, Higham RC. Early Evidence of Safety, Clinical Benefit, and Pharmacokinetics of Roflumilast Cream 0.3% Once Daily for Treatment of Mild or Moderate Plaque Psoriasis in Children Aged 2-11 Years. Pediatr Dermatol. 2026 Jan-Feb;43(1):105-108. doi: 10.1111/pde.70013. Epub 2025 Aug 27. PMID 40862624

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pediatric participants 6-11 years of age were enrolled at 17 study sites in the United States, Canada, and the Dominican Republic.
Groups:
- ARQ-151 Cream 0.3%: Participants apply ARQ-151 cream 0.3% to chronic plaque psoriasis lesions once daily for 4 weeks
Period: Overall Study
Arm/Group | ARQ-151 Cream 0.3%
Started | 20
Completed (Seven of the 20 participants who completed the study are continuing in study ARQ-151-306.) | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ARQ-151 Cream 0.3%
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.8 (1.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of ARQ-151 Cream 0.3%
Description: Plasma levels of circulating roflumilast were determined at 2 points in the study.
Time Frame: Predose on Days 14 and 28
Population: Participants with data available are included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ARQ-151 Cream 0.3%
Number analyzed (Participants) | 18
ng/mL
  Day 14: number analyzed (Participants) | 10
  Day 14 | 3.15 (3.64)
  Day 28 | 1.68 (1.57)

2. Primary Outcome: Plasma Concentration of the Roflumilast Major N-oxide Metabolite
Description: Plasma levels of circulating the roflumilast major N-oxide metabolite were determined at 2 points in the study.
Time Frame: Predose on Days 14 and 28
Population: Participants with data available are included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ARQ-151 Cream 0.3%
Number analyzed (Participants) | 18
ng/mL
  Day 14: number analyzed (Participants) | 10
  Day 14 | 28.9 (41.1)
  Day 28 | 15.7 (15.8)

3. Primary Outcome: Number of Participants With ≥1 Adverse Event (AE)
Description: The number of participants with adverse events during the treatment period is reported. An AE is any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Time Frame: Up to 28 days
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | ARQ-151 Cream 0.3%
Number analyzed (Participants) | 20
Participants | 4

4. Primary Outcome: Number of Participants With Application Site Reactions
Description: The number of subjects experiencing an application site skin reactions by investigator assessment is reported. The investigator assessed for erythema prior to that day's application of investigational product.
Time Frame: Baseline (Day 1), Day 7, and Day 14
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | ARQ-151 Cream 0.3%
Number analyzed (Participants) | 20
Participants
  Day 1: No erythema | 18
  Day 1: Minimal erythema | 0
  Day 1: Definite erythema | 1
  Day 7: No erythema | 17
  Day 7: Minimal erythema | 3
  Day 7: Definite erythema | 0
  Day 14: No erythema | 19
  Day 14: Minimal erythema | 1
  Day 14: Definite erythema | 0

ADVERSE EVENTS:
Time Frame: Up to 28 days
Description: All treated participants are included.
Arm/Group | ARQ-151 Cream 0.3%
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 4/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARQ-151 Cream 0.3% (N=20)
Candida infection (Infections and infestations) | 1
Application site pain (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Perineal pain (Reproductive system and breast disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Perineal erythema (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is supportive of publishing clinical trial findings. The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT04655313/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT04655313/SAP_001.pdf